CLINICAL TRIAL: NCT04049292
Title: Better and Safer Return to Sport After Anterior Cruciate Ligament Reconstruction
Brief Title: Better and Safer Return to Sport
Acronym: BEAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other); International Olympic Committee (Unknown); Swedish Research Council for Sport Science (Other); Linkoeping University (Other Government); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hege Grindem, Associate professor, Norwegian School of Sport Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1886
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Sport Injury
Keywords: anterior cruciate ligament; return to sport; anterior cruciate ligament reconstruction; rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RTS and rehabilitation tool (Experimental): Six months after ACLR, athletes will commence a standardized RTS assessment. The athlete will follow a standardized, sport-specific progression protocol designed to increase athletic confidence and trust in the knee during sports. Readiness to return to full, unrestricted practice will be determined based on 7 time-based, load-based, clinical and functional criteria. If the athlete fails any of the criteria, he or she will continue to participate in restricted practice. Depending on which of the specific criteria the athlete fails, a targeted treatment plan will be developed. Standardized protocols for effusion management, knee control and strength training will be triggered if the athlete fails the criteria for knee joint effusion, hopping and muscle strength, respectively. The RTS assessment and development of the targeted treatment plan will be repeated every 2 months until the athlete is cleared to RTS, up to a maximum of 12 months after ACLR.
  Interventions: Other: Better and safer return to sport (BEAST)
- Usual care (Active Comparator): Athletes will receive usual care as determined by their treating health care professional
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Better and safer return to sport (BEAST) — The RTS assessment includes a Lachman test, modified stroke test, side hop test, triple hop test, and quadriceps muscle power test. The sport-specific progression plans have 6 participation levels in practice and 6 participation levels in match play. A minimum of 2 weeks and 4 training sessions without pain or effusion must be completed before the athlete progresses to the next level. Criteria for full, unrestricted participation in practice: (1)at least 9 months from ACLR, (2)modified stroke test grade 0, (3)completed previous levels in the sport-specific progression plan, (4)negative Lachman test, (5)side hop test limb symmetry at least 90%, (6)triple hop test limb symmetry at least 90%, (7)quadriceps power symmetry at least 90%. The strength training and knee control exercise protocols each have 3-4 different exercises of 3-4 sets that are performed 3 days per week.
  Arms: RTS and rehabilitation tool
Other: Usual care — Usual care is determined by the treating health care professional
  Arms: Usual care

SUMMARY:
A prospective cohort design will be used to assess differences in outcomes between pivoting sport athletes with anterior cruciate ligament reconstruction (ACLR) who follow usual care and those who follow a treatment algorithm with a RTS and rehabilitation tool. Athletes aged 15-40 at injury with primary ACLR who express a goal to return to sports with frequent pivoting are eligible. The RTS and rehabilitation tool includes standardized clinical, functional and muscle strength testing 6, 8, 10, and 12 months after surgery. Individual test results guide progression in sports participation and the content of further rehabilitation according to a standardized algorithm.

DETAILED DESCRIPTION:
Fewer than half of athletes with ACLR return to competitive sports, and, for those who return, 1 in 5 sustain reinjury. Insufficient functional recovery and poor psychological readiness to RTS are thought to contribute to these low RTS rates and high reinjury rates. Previous research has shown that return to sport (RTS) should be delayed until the athlete passes the criteria of a clinical decision-making tool for RTS. However, to successfully improve RTS and reinjury outcomes, it is imperative that a decision-making tool (1) guides RTS decisions at a specific point in time, and (2) directs the planning and execution of treatments that eventually enable the athlete to safely RTS.

Nonprofessional athletes are often discharged from rehabilitation prior to RTS, and most are treated by rehabilitation clinicians who do not have access to the sophisticated and expensive test equipment used in previous research on functional readiness for RTS. The RTS and rehabilitation tool is therefore designed in collaboration with athletes, coaches and primary care physical therapists as a low-cost intervention that is feasible to implement on a broad scale.

The athletes who follow the RTS and rehabilitation tool will be recruited from Oslo, Norway, while the control group that receives usual care will be recruited from the Swedish Knee Ligament register (SPARX study Dnr 2019-04546).

Predefined adjustment factors for the comparative analyses are: age, sex, specific preinjury sport, family history of ACL injury, time from injury to surgery, meniscal and cartilage injury at ACLR, meniscal repair, and ACL graft type. The analysis of reinjury will be adjusted for sports exposure.

Objectives

* To compare 1 and 2-year sports participation, psychological readiness to RTS, knee function and reinjury outcomes between athletes with ACLR who follow a treatment algorithm with a RTS and rehabilitation tool and those who follow usual care
* To assess adherence and barriers to adherence in athletes with ACLR who follow a treatment algorithm with a RTS and rehabilitation tool

ELIGIBILITY:
Inclusion Criteria:

* primary anterior cruciate ligament reconstruction 6 months ago (+- 2 weeks)
* age 15-40 years at the time of anterior cruciate ligament injury
* preinjury participation in level I pivoting sport at least 2 times per week
* expressed goal to return to level I sport

Exclusion Criteria:

* grade 3 injury to the medial collateral ligament, lateral collateral ligament, or posterior cruciate ligament
* contralateral ACL tear
* inability to understand the native language in the country of recruitment
* other serious injury or illness that impairs function
* has access to specialist sports medicine care (e.g., health support from national team) not accessible to all athletes
* derives primary income from sports participation
* member of sports health team present at the majority of the team's training sessions

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Return to sport | 2 years after ACLR
  Participation in preinjury sport (yes/no)
Reinjury | 2 years after ACLR
  Injury to the ACL, medial or lateral meniscus in the ipsi- and contralateral knee (yes/no)

SECONDARY OUTCOMES:
International knee documentation committee subjective knee form | 2 years after ACLR
  Patient-reported measure of knee symptoms, function and activity level, scored 0-100
Anterior cruciate ligament return to sport after injury | 2 years after ACLR
  Patient-reported measure of emotions, confidence in performance, and risk appraisal in relation to RTS, scored 0-100
Adherence/fidelity to the intervention | Monthly self-report 7-14 months after ACLR
  Project-specific questionnaire
Barriers and motivating factors for adherence to the intervention | 14 months after ACLR
  Self-reported on a project-specific questionnaire

OTHER OUTCOMES:
Sports participation | 2 years after ACLR
  Self-reported participation in all sports/physical activity
OSTRC overuse injury questionnaire | 2 years after ACLR
  Oslo Sport Trauma Research Center overuse injury questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hege Grindem, PT PhD, Principal Investigator — Norwegian School of Sport Sciences
Locations (2):
- Norway (2):
  - Norsk Idrettsmedisinsk Institutt, Oslo
  - Idrettens helsesenter, Oslo

IPD SHARING:
Plan to Share IPD: No